CLINICAL TRIAL: NCT03262948
Title: The Randomized,Open, Multicenter Phase III Study to Compare the Effectiveness and Safety of Nab-Paclitaxel Versus Paclitaxel Plus Carboplatin First-Line Therapy Advanced Non Small Cell Lung Cancer Squamous Cell Carcinoma
Brief Title: Nab-Paclitaxel Versus Paclitaxel Plus Carboplatin in Advanced Squamous Cell Non Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NABP201706
Record Dates: First submitted 2017-08-15; First posted 2017-08-28 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 130-nm albumin-bound paclitaxel; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nab-paclitaxel plus carboplatin (Experimental): nab-paclitaxel 260mg/m2,i.v., plus carboplatin AUC = 6,i.v., starting from randomization, once every 3 weeks, for 4-6 cycles, or progression, or intolerance,or death or start a new anti-tumor treatment, whichever occurs first.
  Interventions: Drug: nab-paclitaxel; Drug: Carboplatin
- Paclitaxel plus carboplatin (Active Comparator): paclitaxel 175 mg/m2,i.v., plus carboplatin AUC = 6,i.v., starting from randomization, once every 3 weeks, for 4-6 cycles, or progression, or intolerance,or death or start a new anti-tumor treatment, whichever occurs first.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: nab-paclitaxel — albumin-bound paclitaxel is 260 mg/m2 intravenously over 30 minutes on Days 1 of each 21-day cycle cycle immediately after albumin-bound paclitaxel
  Other Names: keaili
  Arms: nab-paclitaxel plus carboplatin
Drug: Paclitaxel — paclitaxel is 175 mg/m2 intravenously over 3 hours on Days 1 of each 21-day cycle cycle immediately after paclitaxel
  Other Names: aosu
  Arms: Paclitaxel plus carboplatin
Drug: Carboplatin — carboplatin is administered on Day 1 of each 21-day，followed by paclitaxel or nab-paclitaxel
  Other Names: bobei

SUMMARY:
This is a randomized, multicenter, open, controlled phase III trial. 388 subjects with stage IIIB who were not eligible for radical surgery or radiotherapy, stage IV or recurrent squamous cell NSCLC were enrolled in this study .The subjects will be randomly assigned to one of the two treatment groups at a 1: 1 ratio, and stratified by sex, ECOG physical status, smoking status, disease staging.

DETAILED DESCRIPTION:
Subjects will receive one of two treatment regimens:

Group A: intravenous infusion of paclitaxel (albumin binding) 260 mg/m2, intravenous infusion, carboplatin area under curve （AUC) = 6, intravenous infusion, starting from randomization, once every 3 weeks, for 4-6 cycles,or progression, or intolerance, or deth or start a new anti-tumor treatment, whichever occurs first.

Group B: paclitaxel injection 175 mg/m2, intravenous infusion, carboplatin AUC= 6, intravenous infusion, starting from randomization, once every 3 weeks, for 4-6 cycles, or progression, or intolerance,or death or start a new anti-tumor treatment, whichever occurs first.The primary end point is overall response rate (ORR),the secondary endpoint is progression-free survival (PFS), overall survival (OS), safety and Quality of Life (QOL).

ELIGIBILITY:
Inclusion Criteria:

* Accepted the purpose of the trial, the contents , the predicted efficacy, pharmacological effects and the full explanation of the risk and was understood that the subject had signed the informed consent.
* Subjects had histopathologically or cytologically confirmed NSCLC type of squamous cell carcinoma and were documented; (must be provided without radiotherapy, fixed with formalin, paraffin At least 5 sheets of tumor tissue after embedding)
* Subjects were IIIB who were not suitable for radical surgery or radiotherapy, IV or recurrent NSCLC ; (according to the 7th edition of the International Lung Cancer Research Council (IASLC) classification)
* Subjects who were palliative radiotherapy for bone lesions other than the chest were given the study drug according to CTCAE 4.03 toxicity ≤1
* at least one measurable objective lesions according to RECIST1.1 standard
* ECOG score ≤ 1
* Expected survival time ≥ 3 months
* Subjects are well-behaved, able to undergo treatment and follow-up, and voluntarily comply with this study
* ≥ 18 years old male and female
* The childbearing age subjects must agree to take effective contraceptive measures during the trial; the serum or urine pregnancy test must be negative before 24 hours of the start of chemotherapy
* Women must be non-lactating

Exclusion Criteria:

* There is brain metastases;
* The investigators believe that uncontrolled serious medical illnesses that affect the ability of subjects to receive research programs, such as severe medical illnesses, including severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled high blood pressure, Uncontrolled infections, active peptic ulcers;
* Will hinder the understanding or make informed consent or fill in the questionnaire of dementia, mental state changes or any mental illness;
* Any history of allergic or hypersensitivity to any treatment ingredient;
* In the first 5 years of randomization, there were malignant tumors other than NSCLC, except for the treatment of basal cells or squamous cell skin cancer, localized prostate cancer after radical resection, and ductal carcinoma in situ
* Previously received treatment for advanced/metastatic NSCLC. Note: Allow chemotherapy and radiotherapy to be used as part of neoadjuvant/adjuvant therapy as long as the treatment has ended at least 12 months before the diagnosis of advanced or metastatic disease.
* Received a taxane-based regimen as a neoadjuvant/adjuvant therapy for squamous cell carcinoma ;
* Subjects with ≥2 grade peripheral neuropathy according to CTCAE V 4.03;
* Physical examination and laboratory test results are abnormal ANC：<1.5×109 / L； PLT：<100×109/L； Hb: <90g/L
* Abnormal liver function is defined as:

I) total bilirubin (TBil) level:> normal upper limit (ULN) 1.5 times; II) 2.5 times the rate of aspartate aminotransferase (AST) and alanine aminotransferase (ALT)> ULN, and> 5 times ULN if liver metastases are present

* Definition of renal dysfunction:

Serum creatinine> ULN 1.5 times, or creatinine clearance <50ml/min

* Coagulation function abnormal definition:

International Standardization Ratio (INR)> 1.5 times the ULN, and prothrombin time (PT) or activated partial coagulation Blood enzyme time (aPTT)> ULN 1.5 times, unless the subject is receiving anticoagulant therapy

* Hepatitis B surface antigen positive (HBsAg), and peripheral blood hepatitis B virus DNA (HBV-DNA) titer ≥ 1×103copy number / L of the subjects; if HBsAg positive, and peripheral blood HBV-DNA <1 × 103 copy number / L, if the researchers believe that the subjects in a stable phase of chronic hepatitis B and does not increase the risk of subjects, the subjects eligible to be selected
* Hepatitis C virus (HCV) antibody positive or human immunodeficiency virus (HIV) antibody positive
* need to merge other anti-tumor drug treatment
* Received any other test drug treatment or participated in another interventional clinical trial before 30 days of screening period;
* Researchers think it is not suitable for enrolling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
overall respond rate | overall respond rate will be evaluated every 6 weeks until progression or new anti-cancer therapy initiation, up to 22 months.
  the rate of CR and PR

SECONDARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18 months
  progression free survival
os | From date of randomization until the date of death from any cause,assessed up to 18 months
  overall survival
Quality of life assessment | It will be assessed before the administration of drugs at each first day of the chemotherapy cycle,up to 6 cycles,each cycle is 21 days.
  evaluate the QOL according to Functional Assessment of Cancer Therapy-lung (FACT-L)

CONTACTS AND LOCATIONS:
Overall Officials: li zhang, doctor, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Socinski MA, Bondarenko I, Karaseva NA, Makhson AM, Vynnychenko I, Okamoto I, Hon JK, Hirsh V, Bhar P, Zhang H, Iglesias JL, Renschler MF. Weekly nab-paclitaxel in combination with carboplatin versus solvent-based paclitaxel plus carboplatin as first-line therapy in patients with advanced non-small-cell lung cancer: final results of a phase III trial. J Clin Oncol. 2012 Jun 10;30(17):2055-62. doi: 10.1200/JCO.2011.39.5848. Epub 2012 Apr 30. PMID 22547591